CLINICAL TRIAL: NCT03632811
Title: Adaptation of the Questionnaire "Regarding Patient's Quality of Life With Mastocytosis" in the French Language
Acronym: Mc_QoL
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0303; 2018-A02213-52 (Other: ID-RCB)
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Cutaneous Mastocytosis; Indolent Systemic Mastocytosis
Keywords: cutaneous mastocytosis; indolent systemic mastocytosis; quality of life questionnaire in mastocytosis patient
MeSH Terms: conditions — Mastocytosis, Cutaneous; Mastocytosis, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A structured interview with every patient — The comprehension test will be done through structured interviews in which the principal investigator will ask if the patient has had difficulty understanding the recommendations and questions, will check the interpretation of all items and the understanding of each word by the patient. In case of problems, the investigator will propose and / or test translation alternatives, or will ask the patient to propose alternatives.

SUMMARY:
Mastocytosis is a heterogeneous rare disease. A 27-item questionnaire to assess the quality of life of patients with cutaneous/ indolent systemic mastocytosis was developed in the German language and validated in the English language in 2015.

The team of the University Charité Berlin and the company Moxie - intellectual proprietor of the questionnaire - proposed the use of the recommendations of Baiardini et al. 2010, for linguistic adaptation of this questionnaire in other languages.

DETAILED DESCRIPTION:
The first two steps of the program of linguistic translation have already been carried out under the direction and supervision of teams from Charité University, Berlin and Moxie Company. The result of these two steps is a secondary version of the Mc-QoL questionnaire in French. The last step of this adaptation process in the target language (French, France) needs to be carried out and it is the subject of this study.

The objective of this study is the French language adaptation of the Mc-QoL questionnaire in adult patients with indolent cutaneous and / or indolent systemic mastocytosis.

During this study, the second version of the Mc-QoL questionnaire in French will be evaluated on 10 adult patients, with cutaneous and / or indolent systemic mastocytosis and native in the French language. The comprehension tests will be carried out by means of the structured interviews during which the investigator will ask if the patient has had difficulties to understand the recommendations, the questionnaires, will verify the interpretation of all the items and the understanding of each word by the patient. In case of problems, the investigator will propose and / or test translation alternatives, or will ask the patient to propose alternatives.

Revisions to the second version of the Mc-QoL questionnaire in French will be done to rectify the problems identified in the conceptual equivalence. The result will be a third French version of the Mc-QoL questionnaire, which will be the final version.

A report on the interviews will be written in English: it will describe the number of respondents, their age, the time required to complete the questionnaire, the difficulties encountered, the solutions suggested and retained and how the third version of the questionnaire was produced.

ELIGIBILITY:
Inclusion Criteria:

* Adult, native French patient with cutaneous or indolent systemic mastocytosis and follow-up at CEREMAST, Toulouse
* Patient having given his agreement of non-opposition

Exclusion Criteria:

* Minor patient
* Patient with other forms of mast cell pathology except cutaneous and / or indolent systemic mastocytosis
* Patient with no mast cell pathology
* French non-native patient
* Patient in detention or under guardianship
* Patient not affiliated with Social Security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who has indolent cutaneous or systemic mastocytosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
The understanding of aspects of the questionnaire Mc-QoL | 1 day
  The understanding of aspects of the questionnaire Mc-QoL (version "secondary" in French) will be evaluated for each patient:
  - the instructions
The understanding of aspects of the questionnaire Mc-QoL | 1 day
  The understanding of aspects of the questionnaire Mc-QoL (version "secondary" in French) will be evaluated for each patient :
  - the questions (items) and the proposed answers
The understanding of aspects of the questionnaire Mc-QoL | 1 day
  The understanding of aspects of the questionnaire Mc-QoL (version "secondary" in French) will be evaluated for each patient :
  - the layout of the questionnaire
The understanding of aspects of the questionnaire Mc-QoL | 1 day
  The understanding of aspects of the questionnaire Mc-QoL (version "secondary" in French) will be evaluated for each patient :
  - the language (words) used, if it is simple and appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Bulai Livideanu, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No